CLINICAL TRIAL: NCT01715987
Title: A Prospective and Open-Label Study of the Effect on Proximal Tubular Function in Asian-American Patients Receiving Tenofovir Disoproxil Fumarate (TDF) or Entecavir (ETV) for HBV Treatment
Brief Title: Tubular Function in Asian-American Patients Receiving TDF or ETV for HBV Treatment
Status: Terminated | Type: Observational
Sponsor: New Discovery LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: BMS AI463-254
Record Dates: First submitted 2012-10-23; First posted 2012-10-29 (Estimated); Last update posted 2017-09-06 (Actual); Status verified 2015-06

CONDITIONS: Hepatitis B
Keywords: Hepatitis B; Antiviral; Tubular dysfunction; Entecavir; Tenofovir
MeSH Terms: conditions — Hepatitis B | interventions — Tenofovir; entecavir

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood Urine
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Tenofovir Disoproxil Fumarate: Patients who are taking Tenofovir Disoproxil Fumarate.
  Interventions: Drug: Tenofovir Disoproxil Fumarate
- Entecavir: Patients who are taking Entecavir.
  Interventions: Drug: Entecavir

INTERVENTIONS:
Drug: Tenofovir Disoproxil Fumarate — 300mg, oral daily for two years
  Other Names: Viread
  Groups: Tenofovir Disoproxil Fumarate
Drug: Entecavir — 0.5mg oral daily for two years.
  Other Names: Baraclude
  Groups: Entecavir

SUMMARY:
Nucleotide anti-viral analogues, including adefovir and TDF, have demonstrated kidney toxicity in HIV/HBV co-infected patients and HBV mono-infected European patients. Investigators suspected similar kidney proximal tubular injury can also occur in HBV mono infected Asian patients receiving TDF treatment.

DETAILED DESCRIPTION:
The primary objective of this study is to evaluate the safety use of ETV and TDF after at least 144 weeks of treatment in terms of the effects of renal tubular function as determined by (1) 24 hours Urine phosphate (wasting is >1200 mg daily); (2) 24 hours β2-microglobulinuria (NL β2-microglobulin level, <1 mg daily); (3) fractional excretion of uric acid, and (4) fractional tubular reabsorption of phosphorus.

The secondary objectives are to evaluate:

1. To evaluate compare the anti-viral effects of both TDF and ETV as determined the percentage of patient who achieve HBV DNA levels below 60 IU/mL (by quantitative HBV DNA PCR test with lowest level of detection at 60 IU/mL) and ALT normalization by routine biochemical test after 144 weeks of treatment.
2. Serological responses including percentage of patients with HBeAg loss or seroconversion and HBsAg loss or seroconversion with TDF and ETV treatment in Asian-American adults with CHB infection.
3. To evaluate the three-year (one year treatment before enrollment and two year treatment after enrollment) the percentage of patient with anti-HBV drug resistance of TDF and ETV, including genotypic mutations in Asian-American adults with CHB.

ELIGIBILITY:
Inclusion Criteria:

* 18-70 year-old Asian-American male or female patients with HBeAg+ or HBeAg-CHB
* On TDF or ETV mono-therapy for 12-24 months, not previously exposed to other oral HBV drugs, nor received any type of interferon treatment in the past 12 months
* Be willing to participate
* Continuation of HBV treatment is medically indicated. That is for HBeAg-positive subjects, HBeAg remain positive or HBeAg becomes negative but still has detectable DNA by the PCR method; and for HBeAg-negative subjects, HBV DNA is either detectable or undetectable by the PCR method
* No clinical or virologic evidence of anti-HBV resistance to TDF treatment at the time of entering tests
* Serum creatinine < 1.5 mg/L and estimated glomerular filtration rate (creatinine clearance) ≥ 60 mL/min/1.73m2 by the Cockcroft-Gault equation:

  (140-age in years)(body weight [kg] )/((72)(serum creatinine [mg/dl]) ) [Note: multiply estimated rate 0. by 85 for women; use actual body weight]
* Adequate hematologic function (absolute neutrophil count ≥ 1,500/mm3; hemoglobin ≥ 10.0 g/dL)
* To assure all the subjects will be regularly followed per study protocol and minimize the drop off rate, the subjects have to have documented pre-treatment full evaluation and necessary blood tests, medical adherence to HBV treatment, and regular follow-up (i.e., on HBV treatment not missing HBV medication (TDF or ETV) for more than a week, with medical follow-up for HBV treatment at least every 6 month and had all the necessary labs performed.
* In the absence of exclusion criteria.

Exclusion Criteria:

* Ethnicity: Non-Asian CHB patients
* Age: >70 years old
* Body weight and height: BMI ≥ 30
* Concomitant nephrotoxic agents - record all prescription and nonprescription items including herbs and natural remedies, NSAIDs, acyclovir, statins, ACEI or ARBs, Valproate
* Any other antiretroviral meds, antibiotic exposure during study to be noted
* History of HCV, HDV, or HIV co-infection
* Prior history of clinical hepatic decompensation defined as direct (conjugated) bilirubin ≥ 1.2 ULN; PT ≥ 1.2 ULN, platelets ≤ 50,000/mm3, or serum albumin ≤ 3.5 g/dL, ascites, jaundice, encephalopathy, or variceal hemorrhage
* Serum α-fetoprotein ≥ 50 ng/mL
* Evidence of hepatocellular carcinoma (HCC)
* History of solid organ or bone marrow transplantation
* History of malignancies in the past 5 years
* Pregnant women, and women who are breast feeding or who believe they may wish to become pregnant during the course of the study.
* Males and females of reproductive potential who are not willing to use an effective method of contraception during the study. For males, condoms should be used and for females, a barrier contraception method should be used in combination with one other form of contraception.
* History of significant renal disease
* History of significant bone disease
* History of HTN or DM on medical treatment
* Ongoing therapy with any of the following:

  1. Nephrotoxic agents
  2. Parenteral aminoglycoside antibiotics
  3. Cidofovir
  4. Cisplatin
  5. Foscarnet
  6. IV amphotericin B
  7. IV pentamidine
  8. Oral or IV ganciclovir
  9. Cyclosporine
  10. Tacrolimus
  11. IV vancomycin
  12. Chronic daily non-steroidal anti-inflammatory drug therapy
  13. Competitors of renal excretion Systemic chemotherapeutic agents
  14. Systemic corticosteroids
  15. Interleukin-2 (IL-2) and other immunomodulating agents
* Investigational agents (except with the expressed approval of the lead investigators) Administration of any of the above medications must be discontinued at least 30 days prior to the Baseline Visit and for the duration of the study period.

  1. Known hypersensitivity to the study drugs, the metabolites or formulation excipients
  2. Any other condition (including alcohol or substance abuse) or prior therapy that, in the opinion of the Investigators, would make the subject unsuitable for the study or unable to comply with dosing requirements

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Asian Americans with hepatitis B taking Entecavir or Tenofovir.
Sampling Method: Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2012-10; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
renal tubular dysfunction | at 144 week after treatment with antiviral
  renal tubular dysfunction as determined by (1) 24 hours Urine phosphate (wasting is >1200 mg daily); (2) 24 hours β2-microglobulinuria (NL β2-microglobulin level, <1 mg daily); (3) fractional excretion of uric acid, and (4) fractional tubular reabsorption of phosphorus.

CONTACTS AND LOCATIONS:
Overall Officials: Calvin Q Pan, M.D., Principal Investigator — Mount Sinai School of Medicine, New York
Locations (2):
- United States (2):
  - Asian Pacific Liver Center at St. Vincent Medical Center, Los Angeles, California
  - New Discovery LLC, New York, New York